CLINICAL TRIAL: NCT05412953
Title: Tonation Breathing Technique, a Non-Pharmacogenic Method to Ease Aromatase Inhibitor-Induced Musculoskeletal Symptoms - A Pilot Study
Brief Title: Tonation Breathing Technique Method to Ease Aromatase Inhibitor-induced Joint and/or Muscle Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-012300; NCI-2022-01372 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2022-06-03; First posted 2022-06-09 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8
MeSH Terms: interventions — Respiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive care (tonation breathing techniques, questionnaire) (Experimental): Patients participate in tonation breathing techniques twice daily (or more if pain occurs) for 2 weeks. Patients also complete questionnaire at baseline and at 2 weeks.
  Interventions: Other: Questionnaire Administration; Behavioral: Tonation Breathing Technique

INTERVENTIONS:
Other: Questionnaire Administration — Complete questionnaire
Behavioral: Tonation Breathing Technique — Participate in tonation breathing techniques
  Other Names: Breathing and Tonation Technique; TBT

SUMMARY:
This clinical trial evaluates how well tonation breathing techniques (use of a breathing and tonation [creating sounds]) works to ease pain joint and/or muscle pain in patients with stage I-III breast cancer and currently take an aromatase inhibitor. Tonation breathing techniques may help relieve pain in patients with stage I-III breast cancer who are receiving aromatase inhibitor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To study impact of active participation of patients in producing tones in combination with breathing technique, i.e., tonation breathing techniques (TBT) to reduce aromatase inhibitor induced musculoskeletal symptoms.

OUTLINE:

Patients participate in tonation breathing techniques twice daily (or more if pain occurs) for 2 weeks. Patients also complete questionnaire at baseline and at 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Females with stage I-III breast cancer taking adjuvant aromatase inhibitor (AI) (either standard dose of anastrozole 1 mg daily or letrozole 2.5 mg daily or exemestane 25 mg daily) for greater than 30 days experiencing AI induced musculoskeletal pain scores of 5 or higher on a Likert scale will be enrolled
* Subjects should have completed any planned surgery for breast cancer, chemotherapy and radiation therapy at least 30 days prior to enrollment
* Patients should have an Eastern Cooperative Oncology Group (ECOG) performance score of 0-2
* Patients should be at least 18 years old with no maximum age limit

Exclusion Criteria:

* Patients should not have significant underlying pulmonary disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-02-22 (Actual); Primary Completion 2024-06-27 (Actual); Study Completion 2024-06-27 (Actual)

PRIMARY OUTCOMES:
Change in aromatase inhibitor induced musculoskeletal pain symptoms | Baseline to 2 weeks
  Patients will be asked to complete a validated brief pain inventory- SF ( BPI-SF) at baseline and after 2 weeks which would be end of study. The BPI- SF measures pain intensity at its worse in the last week, at its least in the last week in addition to average pain and location of pain. It also measures relief of pain from pain treatments or medications and percentage of relief.

CONTACTS AND LOCATIONS:
Overall Officials: Prema P Peethambaram, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials